CLINICAL TRIAL: NCT02620839
Title: A Phase Ib, Open-label Study of Alpelisib (BYL719) in Combination With Cisplatin in Patients With HPV+ Solid Tumor Malignancies
Brief Title: Phase Ib Study of Alpelisib With Cisplatin in Patients With HPV+ Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Pamela Munster (Other)
Responsible Party: Sponsor-Investigator, Pamela Munster, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 159516; NCI-2017-01680 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumors
Keywords: CDKN2A-p16 Positive; Locally Advanced Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Alpelisib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1A (Experimental): Alpelisib: 200 mg/day, orally, days 1-21 Cisplatin: 30 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin
- Cohort 2A (Experimental): Alpelisib: 250 mg/day, orally, days 1-21 Cisplatin: 30 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin
- Cohort 2B (Experimental): Alpelisib: 250 mg/day, orally, days 1-21 Cisplatin: 35 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin
- Cohort 3A (Experimental): Alpelisib: 300 mg/day, orally, days 1-21 Cisplatin: 30 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin
- Cohort 3B (Experimental): Alpelisib: 300 mg/day, orally, days 1-21 Cisplatin: 35 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin
- Cohort 4A (Experimental): Alpelisib: 350 mg/day, orally, days 1-21 Cisplatin: 30 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin
- Cohort 4B (Experimental): Alpelisib: 350 mg/day, orally, days 1-21 Cisplatin: 35 mg/m^2, intravenously, days 1, 8, 15
  Interventions: Drug: Alpelisib; Drug: Cisplatin

INTERVENTIONS:
Drug: Alpelisib — Given PO
Drug: Cisplatin — Given IV

SUMMARY:
This phase Ib trial studies the best dose and side effects of alpelisib and cisplatin in treating patients with human papillomavirus (HPV) positive solid tumor malignancies. Alpelisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving alpelisib and cisplatin may work better in treating patients with solid tumor malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose and recommended phase 2 dose of alpelisib in combination with weekly cisplatin.

SECONDARY OBJECTIVES:

I. To determine the objective response rate and median progression-free survival with the treatment combination in HPV positive (+) solid tumor malignancies.

II. To characterize the safety profile of the combination.

OUTLINE: This is a dose escalation study.

Patients receive alpelisib orally (PO) once daily (QD) on days 1-14 or 1-21, and cisplatin intravenously (IV) over 1-2 hours on days 1 and 8, or days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign the informed consent form, and able to comply with the study visit schedule and other protocol requirements. Written informed consent obtained prior to any screening procedures.
* Age ≥ 18 years.
* Dose escalation:
* Any locally advanced or metastatic solid tumor malignancy with no curative treatment options available
* Dose expansion:
* HPV-associated locally advanced or metastatic platinum-resistant solid tumor malignancy. HPV positivity defined by positive p16 immunohistochemistry or in-situ hybridization assessment of archival tissue (primary or metastatic) in a CLIA-certified laboratory. Availability of pathology report from CLIA-certified lab demonstrating positive HPV status by p16 IHC or in situ hybridization qualifies for eligibility determination. Analysis of fresh tumor tissue is permitted in cases where archival tissue is not available.
* Platinum resistance defined as prior progression (radiographic or clinical) either during or within 6 months following completion of platinum-based chemotherapy.
* Platinum-based therapy as most recent systemic therapy prior to enrollment allowed but not required
* Patients may have received any number of lines of prior systemic therapy for locally advanced/metastatic disease.
* Eastern Cooperative Oncology Group performance status ≤ 1
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:
* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine < 1.5 x ULN OR Estimated GFR by Cockroft-Gault equation OR 24 hour urine collection ≥ 60 ml/min
* Total serum bilirubin ≤ 1.5 x ULN (< 3 x ULN in patients with documented/suspected Gilbert's disease with concomitant direct bilirubin ≤ 1.5 x ULN)
* Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 x ULN (or ≤ 5 x ULN if liver metastases are present)
* Fasting plasma glucose (FPG) ≤ 140mg/dL or 7.8 mmol/L
* Hemoglobin A1c < 7%
* Patient is able to swallow oral medications.
* Measurable or evaluable disease by RECIST 1.1 in dose escalation. Measurable disease by RECIST 1.1 is required in dose expansion.
* Recovery from all AEs of previous anti-cancer therapies, including surgery, chemotherapy and radiotherapy, to baseline or to CTCAE Grade ≤ 1, except for alopecia.

Exclusion Criteria:

* Prior treatment with PI3K-inhibitor.
* Prior known hypersensitivity to any of the excipients of alpelisib.
* Grade ≥ 2 peripheral neuropathy.
* Grade ≥ sensorineural hearing loss.
* Patients with uncontrolled CNS metastatic involvement. However, patients with metastatic CNS tumors may participate in this study if the patient is:
* > 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
* Clinically stable with respect to the CNS tumor at the time of screening
* Not receiving steroid therapy
* Not receiving anti-convulsive medications that were started for brain metastases.
* Patients who have received prior systemic anti-cancer treatment within 4 weeks or 5 half-lives of prior to starting study treatment, whichever is shorter.
* Prior investigational therapy within 4 weeks of start of study treatment.
* Patients who have received radiotherapy ≤ 2 weeks prior to starting study drugs, with exception of palliative radiotherapy, who have not recovered from side effects of such therapy to baseline or Grade ≤ 1 and/or from whom ≥ 30% of the bone marrow was irradiated.
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study treatment or who have not recovered from side effects of such procedure.
* Clinically significant cardiac disease or impaired cardiac function, such as:
* Congestive heart failure (CHF) requiring treatment (New York Heart Association (NYHA) Grade ≥ 2) or left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
* History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high- grade/complete AV-blockage
* Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft [CABG], coronary angioplasty, or stenting), < 3 months prior to screening
* QT interval adjusted according to Fredericia (QTcF) > 480 msec on screening ECG
* Patients with diabetes mellitus requiring insulin treatment or uncontrolled steroid-induced diabetes mellitus.
* Any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, social/psychological complications.
* Impaired GI function or GI disease that may significantly alter the absorption of oral alpelisib (e.g. Uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or significant small bowel resection).
* Patients who are currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug treatment. A list of prohibited drugs with a known risk of TdP is provided in Appendix.
* Patient is currently receiving treatment with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the start of treatment. Switching to a different medication is allowed. (Refer to Appendix)
* Known positive serology for human immunodeficiency virus (HIV) (baseline testing not required)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
* Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

Sexually active males should use a condom during intercourse while taking drug and for 16 weeks after the final dose of study treatment and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 16 weeks after the final dose of study treatment. Highly effective contraception is defined as either:

Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.

Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study subjects, the vasectomized male partner should be the sole partner for that patient].

Use a combination of the following (both a+b):

Placement of an intrauterine device (IUD) or intrauterine system (IUS) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

For women with therapy-induced amenorrhea, oophorectomy or serial measurements of FSH and/or estradiol are needed to ensure postmenopausal status.

NOTE: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose of alpelisib in combination with cisplatin, based upon evaluation of dose-limiting toxicities and adverse events | Up to 21 days
  Measured using CTCAE v.4.03
Recommended phase 2 dose of alpelisib in combination with cisplatin, based upon evaluation of dose-limiting toxicities | Up to 30 days after the last administration of the study treatment
  Measured using CTCAE v.4.03

SECONDARY OUTCOMES:
Objective Response Rate | Up to 30 days after the last administration of the study treatment
  RECIST v.1.1
Median duration of response | Up to 30 days after the last administration of the study treatment
  RECIST v.1.1
Median Progression-Free Survival | Up to 30 days after the last administration of the study treatment
  RECIST v.1.1
Incidence of adverse events of the treatment combination | Up to 30 days after the last administration of the study treatment
  CTCAE v.4.03

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States